CLINICAL TRIAL: NCT07016113
Title: Comparison of the Effectiveness Between a Combination of 0.005% Latanoprost Gel With 308 nm Excimer Phototherapy and a Combination of 0.1% Mometasone Furoate Cream With 308 nm Excimer Phototherapy on Repigmentation of Nonsegmental Vitiligo in Children
Brief Title: 0.005% Latanoprost Gel for Nonsegmental Vitiligo
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DV-202506.01
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Vitiligo - Macular Depigmentation
Keywords: Latanoprost; Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: Group A: 0.005% latanoprost gel and 308 nm excimer phototherapy Group B: 0.1% mometasone furoate cream and 308 nm excimer phototherapy
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: 0.005% latanoprost gel and 308 nm excimer phototherapy (Experimental): * Apply 0.005% latanoprost gel to the predetermined skin lesions twice daily (morning and evening) every day for 12 weeks.
  * Phototherapy is administered at a dose based on the lesion's location and the response to previous phototherapy sessions. Phototherapy is performed twice a week for 12 weeks.
  Interventions: Drug: 0.005% latanoprost gel
- Group B : 0.1% mometasone furoate cream and 308 nm excimer phototherapy (Active Comparator): * Apply 0.1% mometasone furoate cream to the predetermined skin lesions twice daily (morning and evening) for 12 weeks.
  * Phototherapy is administered at a dose based on the lesion's location and the response to previous phototherapy sessions. Phototherapy is performed twice a week for 12 weeks.
  Interventions: Drug: 0.1% mometasone furoate cream

INTERVENTIONS:
Drug: 0.005% latanoprost gel — - Apply 0.005% latanoprost gel to the predetermined skin lesions twice daily (morning and evening) every day for 12 weeks. - Phototherapy is administered at a dose based on the lesion's location and the response to previous phototherapy sessions. Phototherapy is performed twice a week for 12 weeks.
  Arms: Group A: 0.005% latanoprost gel and 308 nm excimer phototherapy
Drug: 0.1% mometasone furoate cream — - Apply 0.1% mometasone furoate cream to the predetermined skin lesions twice daily (morning and evening) for 12 weeks. - Phototherapy is administered at a dose based on the lesion's location and the response to previous phototherapy sessions. Phototherapy is performed twice a week for 12 weeks.
  Arms: Group B : 0.1% mometasone furoate cream and 308 nm excimer phototherapy

SUMMARY:
Latanoprost, a prostaglandin F2α (PGF2α) analog used for glaucoma treatment, is known to cause iris darkening, hypertrichosis, and periocular skin hyperpigmentation. PGF2α has been shown to stimulate the growth of melanocyte dendrites, increasing dendricity even at low doses, as well as enhancing tyrosinase activity and quantity, thereby promoting repigmentation. Studies on the use of 0.005% latanoprost gel in both children and adults with vitiligo have demonstrated effective repigmentation without reported side effects.

DETAILED DESCRIPTION:
Vitiligo is an acquired pigmentation disorder caused by the progressive loss of melanocytes in the epidermal layer of the skin and/or mucosa, characterized by macules or patches of depigmentation. Vitiligo can occur at any age, including in childhood. Treatment options for vitiligo include medical therapies (topical, systemic, and radiation) as well as surgical approaches. A combination of topical corticosteroids and phototherapy has shown fairly good repigmentation success in treating vitiligo in children. However, long-term use can lead to side effects such as skin atrophy, striae, telangiectasia, hypopigmentation, acneiform eruptions, and hypertrichosis. Latanoprost, a prostaglandin F2α (PGF2α) analog used for glaucoma treatment, is known to cause iris darkening, hypertrichosis, and periocular skin hyperpigmentation. Because of these effects, it has been studied as a treatment for alopecia and hypopigmentation disorders. PGF2α has been shown to stimulate the growth of melanocyte dendrites, increasing dendricity even at low doses, as well as enhancing tyrosinase activity and quantity, thereby promoting repigmentation. Studies on the use of 0.005% latanoprost gel in both children and adults with vitiligo have demonstrated effective repigmentation without reported side effects. To date, there have been no published studies in Indonesia investigating the use of 0.005% topical latanoprost gel for the repigmentation of stable vitiligo lesions in children. Therefore, research comparing the effectiveness of latanoprost gel and 0.1% mometasone furoate cream in combination with phototherapy-the mainstay treatment for pediatric vitiligo in Indonesia-is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo.
* Patients with stable vitiligo for at least 6 months based on the Vitiligo Disease Activity (VIDA) score.
* Aged 10-17 years.
* Affected area <10%.
* Having at least two lesions to be treated. The vitiligo lesions selected for treatment must meet the following criteria:

  1. Relatively the same size, ranging from a minimum of 1 cm² to 4 cm².
  2. Bilateral location on both sides of the body.
  3. A minimum distance of 5 cm between the studied lesions and other vitiligo lesions.
  4. Not located on the palms, soles, or genital area.

Exclusion Criteria:

* Use of topical therapy (corticosteroids, calcineurin inhibitors, psoralen, and antioxidants) for at least 2 weeks before the study, systemic therapy (corticosteroids, antioxidants, and vitamin D) for at least 4 weeks before the study, and phototherapy for at least 4 weeks before the study.
* Presence of other active autoimmune diseases such as type 1 diabetes mellitus, thyroid disease, alopecia areata, rheumatoid arthritis, or Addison's disease, based on medical history and physical examination.
* History of or current skin cancer, photosensitivity, or undergoing radiotherapy.
* Allergy or contraindication to topical corticosteroids or latanoprost.
* History of hypertension, asthma, diabetes mellitus, anemia, kidney, liver, neurological, or cardiovascular diseases.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Area of repigmentation | From enrollment to the end of treatment at 12 weeks
  The percentage level of repigmentation area in lesions before and after therapy.
  Evaluated by Software ImageJ on the week 2, week 4, week 6, week 8, week 10, week 12.
  The assessment categories are as follows: Poor for less than 50%, Fair for 50 to 74%, Good for 75 to 89%, and Excellent for 90 to 100%. These percentage ranges help classify the level of achievement or effectiveness in the evaluation.
Pattern of repigmentation | From enrollment to the end of treatment at 12 weeks
  The pattern of skin color return, such as perifolicular, diffuse, marginal or mixed.
  Evaluated by dermoscopy on the week 2, week 4, week 6, week 8, week 10, week 12.
Number of lesions with repigmentation | From enrollment to the end of treatment at 12 weeks
  The initial appearance of repigmentation on VNS lesions after treatment. Evaluated by dermoscopy on the week 2, week 4, week 6, week 8, week 10, week 12.

SECONDARY OUTCOMES:
VASI score assessment | From enrollment to the end of treatment at 12 weeks
  An assessment to measure the area of depigmented lesions and the severity of depigmentation.
  Evaluated by VASI score on the week 2, week 4, week 6, week 8, week 10, week 12.
  The improvement levels are categorized as follows: Minimal improvement ranges from 0 to +10, Improvement ranges from +10 to 25, Significant improvement ranges from +25 to 50, and Excellent improvement is above +50. These categories help to describe the degree of progress observed.
Side effects and subjective complaints | From enrollment to the end of treatment at 12 weeks
  Side effects and subjective complaints after the intervention. Evaluated by history taking, on the week 2, week 4, week 6, week 8, week 10, and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Reiva F Dwiyana, MD, PhD, Principal Investigator — Hasan Sadikin General Hospital
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

REFERENCES:
- [Result] Anbar TS, El-Ammawi TS, Barakat M, Fawzy A. Skin pigmentation after NB-UVB and three analogues of prostaglandin F(2alpha) in guinea pigs: a comparative study. J Eur Acad Dermatol Venereol. 2010 Jan;24(1):28-31. doi: 10.1111/j.1468-3083.2009.03346.x. Epub 2009 Jul 13. PMID 19627411
- [Result] Korobko IV, Lomonosov KM. A pilot comparative study of topical latanoprost and tacrolimus in combination with narrow-band ultraviolet B phototherapy and microneedling for the treatment of nonsegmental vitiligo. Dermatol Ther. 2016 Nov;29(6):437-441. doi: 10.1111/dth.12383. Epub 2016 Jun 21. PMID 27329330
- [Result] Anbar TS, El-Ammawi TS, Abdel-Rahman AT, Hanna MR. The effect of latanoprost on vitiligo: a preliminary comparative study. Int J Dermatol. 2015;54(5):587-93. doi: 10.1111/ijd.12631. Epub 2014 Dec 29. PMID 25545321
- [Result] Nowroozpoor Dailami K, Hosseini A, Rahmatpour Rokni G, Saeedi M, Morteza-Semnani K, Sadeghi Z, Ghasemzadeh Diva SM, Goldust M, Lotti T, Vojvodic A, Goren A, Sonthalia S, Rathod D. Efficacy of topical latanoprost in the treatment of eyelid vitiligo: A randomized, double-blind clinical trial study. Dermatol Ther. 2020 Jan;33(1):e13175. doi: 10.1111/dth.13175. Epub 2019 Dec 26. PMID 31758835